CLINICAL TRIAL: NCT01406639
Title: Ranibizumab for the Management of Recurrent Epistaxis in Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Ranibizumab for the Management of Recurrent Nosebleeds in Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn due to lack of study population.
Sponsor: University of California, San Diego (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Terence Davidson, Associate Dean/Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091219
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT); Nosebleeds
Keywords: Hereditary Hemorrhagic Telangiectasia (HHT); Nosebleeds; Ranibizumab; Lucentis
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Experimental): Patients treated with topical ranibizumab.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Patients will be treated with a total of 4 applications of ranibizumab in a fine mist spray. This will be done with 2 mgs in 0.2cc; 0.1cc sprayed into each nostril a day; therefore 8 mgs will require 4 days of application. If, following the first treatments, they experience recurrent bleeding (equal to or less than a 75% reduction in their ESS number as compared to pre treatment), they will be offered the opportunity to be prescribed a second administration, to be completed in the same way (4 applications of 4 mg in 0.4 cc with 0.2cc per nostril).
  Other Names: Lucentis

SUMMARY:
This study is for patients with recurrent epistaxis (nosebleeds) as a result of Hereditary Hemorrhagic Telangiectasia (HHT). The aim is to determine if ranibizumab, topically applied will diminish epistaxis in patients with HHT as measured by the HHT Epistaxis Severity Score (ESS), hematocrit, and hemoglobin and serum ferritin levels.

DETAILED DESCRIPTION:
This is an open-label, Phase I study of intranasal administered ranibizumab in subjects with HHT. Plans are to recruit patients with HHT from the UCSD Nasal Dysfunction Clinic.

Those who come for evaluation and are deemed appropriate for topical ranibizumab without laser will be recruited for this study. Ten (10) consented, enrolled subjects will receive a pulsatile nasal irrigator to clean their nose twice daily. They will complete the initial ESS and have a blood test for Hct, Hgb, serum ferritin, liver function tests, renal function tests and if of child-bearing age, a urine pregnancy test. They will return 1 week later and will then receive intranasal sprays of ranibizumab administered once per week during clinic. Patients will be treated with a total of 4 applications of ranibizumab in a fine mist spray. This will be done with 2 mgs in 0.2cc; 0.1cc sprayed into each nostril a day; therefore 8 mgs will require 4 days of application. If, following the first treatments, they experience recurrent bleeding (equal to or less than a 75% reduction in their ESS number as compared to pre treatment), they will be offered the opportunity to be prescribed a second administration, to be completed in the same way (4 applications of 4 mg in 0.4 cc with 0.2cc per nostril).

At the completion of the treatment, subjects will be observed monthly for examination and ESS until 6 months from the first treatment. At 3 and 6 months laboratory tests will be performed.

ELIGIBILITY:
Inclusion Criteria

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Diagnosed with HHT
* Deemed appropriate for topical Ranibizumab without laser, as determined by severity. For the Ranibizumab to be effective, the spray needs to reach the nasal mucosa. Patients will be instructed in nasal irrigation and will only be treated if they can keep their noses clean.
* Severe patients will presumably not achieve this goal, so subjects will be patients with moderate disease as defined by the epistaxis severity score sheet (Appendix B)

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

* Coagulopathy
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Patients who have had bevacizumab therapy, injection, or spray
* Patients with a known reaction based on macular degeneration treatment
* Patients having received VEGF inhibitors in the last 2 years for the treatment of any ophthalmologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Epistaxis as measured by the HHT Epistaxis Severity Score (ESS), hematocrit, and hemoglobin and serum feritin levels. | Monthly until 6 months from the first treatment.
  Epistaxis will be evaluated on a monthly basis by the HHT Epistaxis Severity Score (ESS), hematocrit, and hemoglobin and serum ferritin levels. This will continue through 6 months after the first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Davidson, M.D., Principal Investigator — UCSD